CLINICAL TRIAL: NCT04287608
Title: Observational Study of Conjunctivitis in the Setting of DUPIXENT® Treatment for Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: R668-AD-1884
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Conjunctivitis; Atopic Dermatitis
MeSH Terms: conditions — Conjunctivitis; Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with qualifying conjunctivitis events
  Interventions: Drug: dupilumab
- Patients with no clinical signs of eye inflammation
  Interventions: Drug: dupilumab

INTERVENTIONS:
Drug: dupilumab — No investigational agents will be provided to study patients, and no specific treatment is required during the study. DUPIXENT®-treated patients will receive DUPIXENT as standard of care for the treatment of their AD, as prescribed by their physician. However, continuous treatment with dupilumab for at least 8 weeks is required as a condition for eligibility.
  Other Names: DUPIXENT®; SAR231893; REGN668

SUMMARY:
The primary objective of the study is to characterize the clinical phenotype(s) of DUPIXENT®-associated conjunctivitis events.

The secondary objectives of the study are to characterize the course of conjunctivitis events during the observation period and collect and assess data on treatment for conjunctivitis events and its effectiveness.

ELIGIBILITY:
Key Inclusion Criteria:

* Treatment with DUPIXENT® for AD (per the current US Prescribing Information) should be ongoing, and have been initiated at least 8 weeks prior to study enrollment. NOTE: A single missed dose in the 8 weeks prior to enrollment is allowed.
* Patients with protocol-specified conjunctivitis events must present with active bilateral conjunctivitis (with or without cornea or eyelid involvement) diagnosed by the ophthalmologist (investigator) which meets all of the following criteria:
* Developed (or significantly worsened) while receiving treatment with DUPIXENT® for AD
* Is clinically significant (eg, moderate-to-severe, extensive, persistent, etc) as determined by the investigator
* There is a suspected causal relationship between DUPIXENT® and conjunctivitis because:
* Conjunctivitis is a new-onset condition or an unusual worsening of a preexisting condition (eg, significantly more severe, more extensive, or more protracted than ever before) AND
* No alternative explanation is more plausible, in the opinion of the investigator
* Reference patients must have AD treated with current ongoing treatment with DUPIXENT® for equal or longer duration as compared to group 1, with no clinical signs of ocular inflammation noted during the entire DUPIXENT® treatment

Key Exclusion Criteria:

* Any known medical, social, or personal limitations that are likely to restrict the patient's ability to undergo study visits and complete study procedures (as assessed by the investigator), including hypersensitivity or other contraindications to the anesthetic eye drops used during the ophthalmological examination.

NOTE: Other protocol defined inclusion/exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll DUPIXENT®-treated patients with protocol-specified conjunctivitis events as well as reference patients with no clinical signs of conjunctivitis. Study participants will be recruited from patients being treated with DUPIXENT® for AD according to US Prescribing Information in the real-world setting, who develop conjunctivitis on treatment. These patients will be recruited with the help of a referral network of dermatologists and other physicians who treat patients with moderate-to-severe AD.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Baseline Ophthalmologist Diagnosis | Initial Visit (Day 1)
  Diagnosis includes: symptoms and morphological features of conjunctivitis
Proportion of patients in each category of ophthalmologist diagnoses | Initial Visit (Day 1)
  Symptoms / Morphological features
Proportion of patients with symptoms | Initial Visit (Day 1) up to week 52
  Symptoms include but are not limited to: infection, dry eye, cytological shifts, etc
Proportion of patients with morphological features | Initial Visit (Day 1) up to week 52
  Morphological features include but are not limited to: bulbar redness, limbal redness, lid redness, lid roughness, etc. and associated conditions may include blepharitis, keratitis, etc.
Proportion of conjunctivitis events by severity | Initial Visit (Day 1) up to week 52
  Severity is based on the nature of the event, intensity of signs and/or symptoms, current functional impairment, and potential long-term health hazards related to the event. 3-point scale: Mild, Moderate or Severe.
Duration of conjunctivitis event(s) in patients whose conjunctivitis resolved | Up to week 52
Proportion of patients with conjunctivitis event resolution | Up to week 52
Proportion of patients who discontinued DUPIXENT® due to conjunctivitis events | Up to week 52
Ophthalmologists assessment of treatment effectiveness, overall and by clinical phenotype based on a 5-point scale. | Up to week 52
  Treatment Effectiveness assessed on a 5-point scale: Poor, Fair, Good, Very Good, Excellent
Change in eosinophil counts and other cells identified by impression cytology from the conjunctival tissue | Up to week 52 or resolution
  Measured by conjunctival impression sample (EyeprimTM) for cytology and RNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (15):
- United States (15):
  - Regeneron Study Site, Irvine, California
  - Regeneron Study Site, Palo Alto, California
  - Regeneron Study Site, Pasadena, California
  - Regeneron Study Site, Miami, Florida
  - Regeneron Study Site, New Orleans, Louisiana
  - Regeneron Study Site, Baltimore, Maryland
  - Regeneron Study Site, Boston, Massachusetts
  - Regeneron Study Site, Great Neck, New York
  - Regeneron Study Site, New York, New York
  - Regeneron Study Site, Portland, Oregon
  - Regeneron Study Site, Philadelphia, Pennsylvania
  - Regeneron Study Site, Pittsburgh, Pennsylvania
  - Regeneron Study Site, Memphis, Tennessee
  - Regeneron Study Site, Dallas, Texas
  - Regeneron Study Site, Houston, Texas

REFERENCES:
- [Derived] Asbell P, Akpek E, Chamberlain W, Chen Z, Lawless E, Van Spall M, Ozturk ZE, Shumel B. Conjunctivitis in Adults with Atopic Dermatitis Treated with Dupilumab: An Observational Study of Clinical Characteristics, Symptomatology, and Treatment. Adv Ther. 2025 Jul;42(7):3285-3305. doi: 10.1007/s12325-025-03209-4. Epub 2025 May 19. PMID 40388089